CLINICAL TRIAL: NCT04235309
Title: Physical Resilience: Indicators and Mechanisms in the Elderly (PRIME) Collaborative Phase 2
Acronym: PRIME-Knee
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00103483; 4UH3AG056925-03 (NIH)
Record Dates: First submitted 2020-01-17; First posted 2020-01-21 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Resilience; Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from study participants at the baseline visit (before surgery) and 24 hours after surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total Knee Replacement Cohort: Any patients who are scheduled to undergo a total knee replacement.

SUMMARY:
The purpose of this study is to examine underlying physical resilience (the ability to bounce back) in response to a specific stressor (total knee replacement).

DETAILED DESCRIPTION:
In general, a person's specific resilience (ability to bounce back from a stressor) is thought to be dependent upon that person's specific biological and genetic makeup. However, these specific elements remain poorly understood. The purpose of this study is to identify important predictors and characteristics of resilience in response to a total knee replacement by examining baseline resilience (prior to surgery) and post-surgical resilience at multiple time points, allowing us to track resilience outcomes over time.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* Ability to speak English
* Planned elective knee replacement orthopedic surgery lasting 2 or more hours and requiring overnight observation or inpatient stay
* Community dwelling

Exclusion Criteria:

* Unable to ambulate independently, with or without assistive device
* Known dementia or screening 3MS score <=77
* Inmate of a correctional facility (i.e. prisoners)
* Active non-skin cancer or medical treatment for non-skin cancer with 12 months (chemotherapy, radiation, immunotherapy, hormonal therapy)
* Vision or hearing impairment that, after best accommodation, prevents reliable cognitive assessment (visual/hearing) and/or precludes telephone interviews (hearing)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prospective observational study of n=250 adults aged 60 years and older undergoing elective total knee replacements with 6 months of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Change in musculoskeletal resiliency following orthopedic surgery as measured by physical activity (step counts) | Baseline, 1 week, 1 month, 2 months, 4 months and 6 months
  As measured by a Garmin device worn by participants
Change in musculoskeletal resiliency following orthopedic surgery as measured by Lower Extremity Physical Activities of Daily Living (LE PADLs) | Baseline, 6 months
  Scores are measured from 0 to 45. Higher scores are associated with more limited LE PADLs.
Change in musculoskeletal resiliency following orthopedic surgery as measured by PROMIS Pain Intensity | Baseline, 1 week, 1 month, 2 months, 4 months and 6 months
  Scores are measured from 3 to 15. Higher scores are associated with more intense pain.
Change in musculoskeletal resiliency following orthopedic surgery as measured by PROMIS Pain Interference | Baseline, 1 week, 1 month, 2 months, 4 months and 6 months
  Scores are measured from 6 to 30. Higher scores are associated with increased pain interference.
Change in cognitive resiliency following orthopedic surgery as measured by 3D-CAM. | Baseline, 1 week
  Scored as positive or negative. Positive indicates the presence of delirium.
Change in cognitive resiliency following orthopedic surgery as measured by cognitive change index (CCI) for patient. | Baseline, 1 month, 2 months, 4 months, 6 months
  Scores range from 20 - 100. Higher scores are associated with increased cognitive decline.
Change in cognitive resiliency following orthopedic surgery as measured by cognitive change index (CCI) for informant about patient. | Baseline, 1 month, 2 months, 4 months, 6 months
  Scores range from 20 - 100. Higher scores are associated with increased cognitive decline.
Change in association between in vitro immune resiliency and resilient outcomes following elective orthopedic surgery. | Baseline, Post-operative Day 1
  Whole blood samples containing PBMCs collected before/after surgery will be challenged with LPS and influenza vaccine to assess the cellular immune response using previously identified biomarkers of resiliency and RNA-seq analysis to identify novel biomarkers and molecular signatures.

SECONDARY OUTCOMES:
Change in dual task gait speed | Baseline, 6 months
  Score of combined walking and verbal fluency test
Change in tissue oxygenation index (TOI) | Baseline, 6 months
  Measured using fNIRs (functional near infrared spectroscopy)
Intraoperative electrocardiography (ECG) RR variability | Surgery up to three hours
  Measured as intra-operative ECG RR intervals collected from the heart monitor

CONTACTS AND LOCATIONS:
Overall Officials: Cathleen S Colon-Emeric, MD, MHS, Principal Investigator — Duke University; Heather E Whitson, MD, MHS, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Regional Hospital, Durham, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No